CLINICAL TRIAL: NCT04185818
Title: Citizen Science: The People's Trial: A Randomised Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National University of Ireland, Galway, Ireland (Other)
Collaborators: Health Research Board, Ireland (Other)
Responsible Party: Principal Investigator, Prof. Declan Devane, Scientific Director, HRB-Trials Methodology Research Network, National University of Ireland, Galway, Ireland
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: HRB.ThePeople'sTrial
Record Dates: First submitted 2019-11-28; First posted 2019-12-04 (Actual); Last update posted 2020-01-31 (Actual); Status verified 2020-01

CONDITIONS: Sleep
Keywords: sleep, book, read, bed
MeSH Terms: conditions — Bornholm Eye Disease

STUDY DESIGN:
Intervention Model Description: The People's Trial is an online pragmatic, randomised controlled trial.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reading group (Experimental): Participants will:
  1. Read a book for 15 to 30 mins
  2. Read immediately before trying to go to sleep.
  Interventions: Other: Reading a book
- Control Group (No Intervention): Participants will:
  1. Not read a book

INTERVENTIONS:
Other: Reading a book — Participants requested to specify usual genre of book they read.
  1. Fiction
  2. Non-Fiction
  3. Other
  4. Don't usually read a book in bed
  Arms: Reading group

SUMMARY:
The People's trial is an online pragmatic, randomised controlled trial to determine if reading a book in bed makes a difference to sleep in comparison to not reading a book in bed.

DETAILED DESCRIPTION:
The People's Trial seeks to help enhance the public's understanding of randomised trials by facilitating the involvement of the public in the trial research process. The public have, through an online format, guided the development and design of The People's Trial randomised controlled trial. The People's trial is a parallel, online randomised controlled trial to determine if reading a book in bed makes a difference to sleep in comparison to not reading a book in bed.

Members of the public will be recruited through online platforms. Informed consent will be obtained from all participants prior to trial registration. Consent forms will be provided online prior to registration for The People's Trial. Participants will be required to acknowledge that they have read the consent form and give consent to proceed with trail registration.

Participants will be randomly allocated into one of two groups:

Group 1: Reading a book in bed

Group 2: Not reading a book in bed

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age on enrollment;
* English speaking;
* ability to read;

Exclusion criteria

* Members of the public who are unwilling or unable to give informed consent.
* Unable to go to bed and wake up at the same time as normal for the study duration.
* Unable to sleep in their own bed, in their own home for the study duration
* Unable to not eat food or drink caffeinated drinks within 1 hour of bed for the study duration

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2019-12-04 (Actual); Primary Completion 2020-02-29 (Estimated); Study Completion 2020-04-01 (Estimated)

PRIMARY OUTCOMES:
Overall sleep quality | From time of randomisation- refers to sleep in the last 7 days only
  Sleep quality will be measured using the single item sleep quality scale (SQS) (Snyder et al 2018). The SQS is a self-administered questionnaire in which respondents rate overall quality of sleep over a 7-day recall period on a discretizing visual analogue scale from 0 to 10 (0 = terrible, 1-3 = poor, 4-6 = fair, 7-9 = good, and 10 = excellent)

SECONDARY OUTCOMES:
Sleep Disturbance | From time of randomisation- refers to sleep in the last 7 days only
  This will be measured using the PROMIS Short Form Sleep Disturbance Scale which measures eight items on 5-point scale to rate the frequency of problems related to insufficient sleep in the past seven days
Daytime sleepiness | From time of randomisation- refers to sleep in the last 7 days only
  Perceptions of daytime sleepiness will be measured using a a single item with a 10-point scale. Respondents are instructed to indicate their sleepiness at that moment by choosing a number between 1 (not sleepy at all) and 10 (very sleepy). Others have found a single item to measure sleep quality produces reproducible and valid data (Cappelleri, et al 2009, Riegel et al 2013).

CONTACTS AND LOCATIONS:
Overall Officials: Declan Devane, Professor, Principal Investigator — National University of Ireland, Galway
Locations (1):
- National University of Ireland Galway, Galway, Co. Galway, Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Finucane E, O'Brien A, Treweek S, Newell J, Das K, Chapman S, Wicks P, Galvin S, Healy P, Biesty L, Gillies K, Noel-Storr A, Gardner H, O'Reilly MF, Devane D. The People's Trial: supporting the public's understanding of randomised trials. Trials. 2022 Mar 9;23(1):205. doi: 10.1186/s13063-021-05984-1. PMID 35264220
- [Derived] Finucane E, O'Brien A, Treweek S, Newell J, Das K, Chapman S, Wicks P, Galvin S, Healy P, Biesty L, Gillies K, Noel-Storr A, Gardner H, O'Reilly MF, Devane D. Does reading a book in bed make a difference to sleep in comparison to not reading a book in bed? The People's Trial-an online, pragmatic, randomised trial. Trials. 2021 Dec 4;22(1):873. doi: 10.1186/s13063-021-05831-3. PMID 34996514